CLINICAL TRIAL: NCT00717106
Title: Observational Study of the Sleuth Implantable ECG Monitoring System
Acronym: OBSERV-ECG
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Transoma Medical (Industry)
Responsible Party: Wim Stegink, Transoma Medical
Other Study IDs: CLP-007
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Syncope; Presyncope; Fainting; Cardiac Arrhythmia
Keywords: ILR; ECG monitoring; cardiac arrhythmia; syncope; presyncope; fainting
MeSH Terms: conditions — Syncope; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to obtain information on real-world device performance clinical assessments and clinical outcomes of patients receiving the Sleuth Implantable ECG Monitoring System.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical syndromes or situations at increased risk of cardiac arrhythmias
* Patients who experience transient symptoms that may suggest a cardiac arrhythmia

Exclusion Criteria:

* Patients that have had a myocardial infarction (MI) < 30 days prior to implant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cardiology or primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2008-07

PRIMARY OUTCOMES:
Time to diagnosis | one year

CONTACTS AND LOCATIONS:
Overall Officials: Wim Stegink, Study Director — Transoma Medical
Locations (8):
- United States (8):
  - Piedmont Hospital, Atlanta, Georgia
  - Western Maryland Health Systems, Cumberland, Maryland
  - Cardiology Consultants of East Michigan, Lapeer, Michigan
  - St. Luke's - Roosevelt, New York, New York
  - SUMMA-NEOCS Health Systems, Akron, Ohio
  - Main Line Health - Lankenau Hospital, Wynnewood, Pennsylvania
  - Center for Cardiac Arrhythmias, Houston, Texas
  - Morgantown Internal Medicine Group, Morgantown, West Virginia